CLINICAL TRIAL: NCT02830971
Title: Effect of Specific Training for Mastery in Doing Different Techniques in Intensive Care Unit: Developing a Standardized Learning Curve
Brief Title: Developing a Standardized Learning Curve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Shahid Beheshti University (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Post doc, PhD, RN, Baqiyatallah Medical Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BUMS Protocl
Record Dates: First submitted 2016-07-04; First posted 2016-07-13 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Registered Nurses; Nursing Personnel; Motor Skills
Keywords: standardized learning curve; Nurse; intensive care unit; Mastery; Training; Developing; Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clinical specific education (Other): Providing clinical skills conditions
  Interventions: Procedure: Doing Different ICU techniques and skills

INTERVENTIONS:
Procedure: Doing Different ICU techniques and skills

SUMMARY:
The nurses were learned the theoretical and practical skills previously during their studentship period. The procedures will be the first time the nurses wanted to perform in ICU. All clinical situations including patient, procedure, and shift will be similar for nurses. The end point will be reaching to the 95 score of learning curve. The reason for selection less than 5 percent variation was the flattening of learning curve (the plateau section).

DETAILED DESCRIPTION:
All new registered nurses in intensive care unit (ICU) from 1 April 2016 until next 24 months from 10 mixed beds ICUs will be selected through convenience sampling and according to fulfilling the inclusion criteria.

For data collection, a specific checklist as many as selected techniques according to the three panel of expert sessions was validated. The members of expert panel were three intensivists, five anesthesiologists, three pulmonologists, five internists, one nephrologist, one cardiologist, and ten highly experienced ICU nurses. Firstly, extensive review of the literature based on the latest documents and articles for techniques was done. The Kendal agreement coefficient between the panel of expert members for selecting the primary materials to constitute the checklist was 0.976 (P Value <0.0001). According to the extensive review of the literature, a primary checklist as many as selected techniques was generated. The primary checklist as many as selected techniques generated in the first expert panel session. After the 90 minutes discussion about the primary checklist as many as selected techniques, the primary consensus was achieved. The primary checklist as many as selected techniques sent to the expert members for purifying, improving and editing. The results of the second 120 minutes distance session were analyzed meticulously by principle investigator and two independent researchers (K=0.943 with P Value <0.0001). Based on the results of the second session, the third version of the checklists as many as selected techniques was prepared. According to the 120 minutes final session, the checklists as many as selected techniques for clinical survey was prepared. The checklists had different domains according to the selected techniques. The scoring of each checklist's questions was based on the 3 status. Ability to perform alone (2 score), ability to perform with helping (1 score) and inability to perform (0 score). Each question had specific importance coefficient among 1 to 5. The philosophy of the different coefficients for the questions in the domains was related to the importance degree of question. Thus, besides the domain scores, each domain had specific importance coefficient. The total score of the checklist comes from multiplying the question score to question importance coefficient with percent. Then, the highest score of the checklist was 100 percent and the lowest score was 0 percent. The nurses received full classical education according to the final three-step checklist components by a full ICU trainer in five 120 minutes sessions as theoretically. The trainer did not inform from the research questions and study. During the three validation sessions, content validity ration (CVR) with 28 panelists were 0.59 and content validity index (CVI) 0.95. Reliability of the checklist was determined based on the inter-rate reliability with Kappa agreement test among principle investigator and intensivists (r= 0.94), anesthesiologists (r= 0.92), pulmonologists (r= 0.90), internists (r= 0.93), nephrologist (r= 0.97), cardiologist (r= 0.95), and three of the nurses (r= 0.91, 90, and 92), separately. Reliability of the checklist was determined based on the intera-rate reliability with Kappa agreement test by principle investigator (r= 0.96), intensivists (r= 0.91), anesthesiologists (r= 0.92), pulmonologists (r= 0.94), internists (r= 0.92), nephrologist (r= 0.93), cardiologist (r= 0.90), and three of the nurses (r= 0.90, 93, and 94), separately. For decreasing the researcher effect on the nurses, the results of two primary weeks will not be considered. Following each nurse will be continued until achieving the flattening of the learning curve.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* nothing already done the technique in ICU
* Not having the preventing physical deformity for doing the skills
* Working as the newly registered nurse in the unit as long as the study is progress

Exclusion Criteria:

* Any situations and conditions will insult the inclusion criteria.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2018-04 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
level of nurse expertise | Six months
  The checklist contained steps for performance skills rated on a 1 to 3 scoring scale (1= The researcher used the checklist to assess the nurse's mastery level while changing a skills and recorded his/her score on the learning curve based on a 0 (no mastery) to 100 (complete mastery) scoring scale.Required Standard frequency for skills performance based on learning curve plateau, achievement of 75% of expertise and, 75 percent of nurses who achieved 75% of expertise in the following skills.

SECONDARY OUTCOMES:
Effect of GPA on the level of nurse expertise | Six months
  The effect of GPA will be measured on the level of nurse expertise

CONTACTS AND LOCATIONS:
Overall Officials: Amir Vahedian-azimi, Postdoc, Principal Investigator — Baqiyatallah Universiy of Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
After the study termination, data will be entered.

REFERENCES:
- [Derived] Vahedian-Azimi A, Rahimi-Bashar F, Pourhoseingholi MA, Salesi M, Shamsizadeh M, Jamialahmadi T, Gohari-Moghadam K, Sahebkar A. Effect of the Specific Training Course for Competency in Doing Arterial Blood Gas Sampling in the Intensive Care Unit: Developing a Standardized Learning Curve according to the Procedure's Time and Socioprofessional Predictors. Biomed Res Int. 2021 Feb 13;2021:2989213. doi: 10.1155/2021/2989213. eCollection 2021. PMID 33628776